CLINICAL TRIAL: NCT04485871
Title: White Adipose Tissue LDL Receptors and Omega-3 as Modulators of the Risk for Type 2 Diabetes in Subjects With Normal Plasma LDL Cholesterol
Brief Title: Targeting Risk Factors for Diabetes in Subjects With Normal Blood Cholesterol Using Omega-3 Fatty Acids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, May Faraj, PDt, PhD, Professor, Institut de Recherches Cliniques de Montreal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-1035; NUT407816 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2020-07-16; First posted 2020-07-24 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Inflammation; Insulin Sensitivity/Resistance; Fatty Acids, Omega-3
Keywords: Proprotein Convertase Subtilisin / kexin Type 9 (PCSK9); NLRP3 inflammasome; Eicosapentaenoic acid (EPA); Docosahexaenoic acid (DHA); White adipose tissue; Fat metabolism; ApoB-lipoproteins; LDL receptors (LDLR); Cluster of differentiation 36 (CD36)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Insulin Resistance; Hypercholesterolemia, Autosomal Dominant, 3; Hyperlipoproteinemia Type II | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Intervention Model Description: Subjects (N=48) will be recruited with the same inclusion/exclusion criteria and will received the same omega-3 intervention. After completion of recruitment, subjects will be stratified into 2 groups (24/group) based on a baseline plasma PCSK9 for group characterisation and comparison.
Masking Description: However, subjects will not know into which group they were stratified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omega-3 fatty acids (Experimental): 3.6 g EPA:DHA / day (2:1)
  Interventions: Dietary Supplement: Omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids — Triple Strength Omega-3 from Webber Naturals; 4 oral softgels (600 mg EPA and 300 mg DHA / softgel)
  Other Names: Triple Strength Omega-3 from Webber Naturals

SUMMARY:
Every 3 minutes a new case of diabetes is diagnosed in Canada, mostly type 2 diabetes (T2D) increasing the risk for heart disease. T2D and heart disease share many common risk factors such as aging, obesity and unhealthy lifestyle.

Paradoxically however, while lowering blood LDL, commonly known as "bad cholesterol", is protective against heart disease, research over the past 10 years have shown that the lower is blood LDL, the higher is the chance of developing T2D. This phenomena is happening whether blood LDL is lowered by a common drug against heart disease called Statins, or by being born with certain variations in genes, some of which are very common (~80% of people have them).

To date, it is unclear why lowering blood LDL is associated with higher risk for diabetes, and whether this can be treated naturally with certain nutrients.

Investigators believe that lowering blood LDL by forcing LDL entry into the body tissue through their receptors promotes T2D. This is because investigators have shown that LDL entry into human fat tissue induces fat tissue dysfunction, which would promote T2D especially in subjects with excess weight.

On the other hand, investigators have shown that omega-3 fatty acids (omega-3) can directly treat the same defects induced by LDL entry into fat tissue. Omega-3 is a unique type of fat that is found mostly in fish oil.

Thus the objectives of this clinical trial to be conducted in 48 subjects with normal blood LDL are to explore if:

1. Subjects with higher LDL receptors and LDL entry into fat tissue have higher risk factors for T2D compared to subjects with lower LDL receptors and LDL entry into fat tissue
2. 6-month supplementation of omega-3 from fish oil can treat subjects with higher LDL receptors and LDL entry into fat tissue reducing their risk for T2D.

This study will thus explore and attempt to treat a new risk factor for T2D using an inexpensive and widely accessible nutraceutical, which would aid in preventing T2D in humans.

DETAILED DESCRIPTION:
Type 2 (T2D) and cardiovascular disease (CVD) share many risk factors, whose accumulation over years lead to disease onset. However, while lowering plasma low-density lipoprotein cholesterol (LDLC) is cardio-protective, novel evidence over the past 10 years established a role for common LDLC-lowering variants and widely used hypocholesterolemic Statins in higher risk for T2D. This diminishes the cardio-protective role of low plasma LDLC. As these conditions decrease plasma LDLC by increasing tissue-uptake of LDL, a role for LDL receptor (LDLR) pathway was proposed. However underlying mechanisms fueling higher risk for T2D with upregulated LDLR pathway, and nutritional approaches to treat them are unclear.

The central hypothesis examined in this trial is that upregulating receptor-mediated uptake of LDL on white adipose tissue provokes the activation of an innate immunity pathway (the Nucleotide-binding domain and Leucine-rich repeat Receptor, containing a Pyrin domain 3 (NLRP3) inflammasome) leading to the accumulation of risk factors for T2D in subjects with normal plasma LDLC. This can be treated by 6-month supplementation of omega-3 fatty acids (omega-3).

To examine this hypothesis in vivo, ex vivo and in vitro, a clinical trial in conjunction with mechanistic basic research studies have been initiated at the Montreal Clinical Research Institute (IRCM). Forty eight volunteers will be recruited through advertisements in French/English newspapers and online (e.g. Google, Facebook) and placed on a 6-month supplementation of 3.6 g omega-3 per day. Participants will be stratified into 2 groups (N=24/group) with higher and lower white adipose tissue surface-expression LDL receptors (LDLR and CD36) using median plasma PCSK9 (Proprotein Convertase Subtilisin/Kexin type 9) per sex. Plasma PSCK9 will be used as investigators have shown that it is negatively associated with white adipose tissue surface-expression of LDLR and CD36.

The duration of this study is about 8 months (33 weeks) divided into 5 parts:

A. Screening and evaluation of eligibility for the study

B. Weight stabilisation (+/- 2 kg change over 4 weeks) and confirmation of eligibility after a medical examination by IRCM physician collaborators.

C. Baseline testing over 2 days (1- 4 weeks apart) to assess participants risk factors for T2D: white adipose tissue NLRP3 inflammasome activity, white adipose tissue physiology and function (ex vivo after a subcutaneous needle biopsy), systemic inflammation, dietary fat clearance (after a high fat meal), and insulin secretion and sensitivity (by gold-standard Botnia clamp technique). Participants will also be phenotyped for body composition (by dual energy x-ray absorptiometry), resting energy expenditure (by indirect calorimetry), dietary intake (by 3-day dietary journals) and physical activity level (by a questionnaire).

D. 24-week intervention with omega-3 fatty acid supplementation (3.6 g eicosapentaenoic acid (EPA) and docosahexaenoic (DHA), 2:1)

E. Post intervention testing starting over 2 days (1- 4 weeks apart) to assess risk factors for T2D that were measured at baseline.

Investigators hypothesize that subjects with low plasma PCSK9 (i.e. with higher white adipose tissue LDLR and CD36) will have higher risk factors for T2D at baseline and that the omega-3 intervention will eliminate group-differences in these risk factors.

ELIGIBILITY:
Inclusion Criteria:

Men and post-menopausal women:

* Having a body mass index (BMI= 25-40 kg/m2)
* Aged between 45 and 74 years
* Having confirmed menopausal status (FSH ≥ 30 U/l)
* Non-smoker
* Sedentary (less than 2 hours of structured physical exercise (ex: sports club) per week)
* Low alcohol consumption: less than 2 alcoholic drinks/day

Exclusion Criteria:

* Plasma LDL cholesterol > 3.5 mmol/L (i.e. > 75th percentile in a Canadian population).
* Elevated risk of cardiovascular disease (≥ 20% of calculated Framingham Risk Score) who would require immediate medical intervention by lipid-lowering agents.
* Prior history of cardiovascular events (like stroke, transient ischemic attack, myocardial infarction, angina, heart failure…)
* Systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg
* Type 1 or 2 diabetes or fasting glucose > 7.0 mmol/L
* Prior history of cancer within the last 3 years
* Thyroid disease - untreated or unstable
* Anemia - Hb < 120 g/L
* Renal dysfunction or plasma creatinine > 100 µmol/L
* Hepatic dysfunction - AST/ALT > 3 times normal limit
* Blood coagulation problems (i.e. bleeding predisposition)
* Autoimmune and chronic inflammatory disease (i.e. celiac, inflammatory bowel, Graves, multiple sclerosis, psoriasis, rheumatoid arthritis, and lupus).Known history of difficulties accessing a vein
* Claustrophobia
* Sleep apnea
* Seizures
* Concomitant medications: Hormone replacement therapy (except thyroid hormone at a stable dose), systemic corticosteroids, anti-psychotic medications and psycho-active medication, anticoagulant or anti-aggregates treatment (Aspirin, NSAIDs, warfarin, coumadin..), adrenergic agonist, anti-hypertensive drugs, weight-loss medication, lipid lowering medication
* Known substance abuse
* Already taking more than 250 mg of omega-3 supplements (EPA/DHA) per day
* Allergy to seafood or fish
* Allergy to Xylocaine
* Unable to eat the components of the high fat meal (croissant, cheese, bacon, brownies)
* None compliance to the study requirements (i.e. not being fasting) or cancellation of the same scheduled testing visit more than once.
* Lack of time to participate in the full length of the study (33 weeks)
* Have exceeded the annual total allowed radiation dose (like X-ray scans and/or tomography in the previous year or in the year to come) according to the physician's judgement.
* All other medical or psychological conditions deemed inappropriate according to the physician

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Fasting white adipose tissue NLRP3 inflammasome activation | Baseline
  White adipose tissue medium accumulation of interleukin 1 beta (IL-1β) ex vivo over 4 hours (pg/mg tissue by AlphaLISA)
Fasting white adipose tissue NLRP3 inflammasome activation | At 24 weeks
  White adipose tissue medium accumulation of interleukin 1 beta (IL-1β) ex vivo over 4 hours (pg/mg tissue by AlphaLISA)

SECONDARY OUTCOMES:
Fasting plasma PCSK9 concentration | Baseline
  Plasma PCSK9 (g/L by ElISA kit)
Fasting plasma PCSK9 concentration | At 24 weeks
  Plasma PCSK9 (g/L by ElISA kit)
White adipose tissue receptors for apoB-lipoproteins | Baseline
  Fasting and 4 hour-postprandial change in white adipose tissue surface-expression LDLR and CD36 (% of control by immunohistochemistry in white adipose tissue slides)
White adipose tissue receptors for apoB-lipoproteins | At 24 weeks
  Fasting and 4 hour-postprandial change in white adipose tissue surface-expression LDLR and CD36 (% of control by immunohistochemistry in white adipose tissue slides)
White adipose tissue inflammation profile | Baseline
  Fasting and 4 hour-postprandial change in NLRP3 inflammasome related inflammatory parameters; including gene expression of IL1B, NLRP3 and ADGRE1 (by RT-PCR) and secretion of IL-1β and IL-1Ra (per mg tissue by AlphaLISA)
White adipose tissue inflammation profile | At 24 weeks
  Fasting and 4 hour-postprandial change in NLRP3 inflammasome related inflammatory parameters; including gene expression of IL1B, NLRP3 and ADGRE1 (by RT-PCR) and secretion of IL-1β and IL-1Ra (per mg tissue by AlphaLISA)
White adipose tissue function ex vivo | Baseline
  Fasting and 4 hour postprandial change in situ lipoprotein lipase activity (nmol 3H-triglyceride/mg tissue)
White adipose tissue function ex vivo | At 24 weeks
  Fasting and 4 hour postprandial change in situ lipoprotein lipase activity (nmol 3H-triglyceride/mg tissue)
Postprandial fat metabolism | Baseline
  Area under the 6 hour time curve of plasma triglycerides (mmol/hour) after a high-fat meal (66% fat)
Postprandial fat metabolism | At 24 week
  Area under the 6 hour time curve of plasma triglycerides (mmol/hour) after a high-fat meal (66% fat)
Systemic inflammation | Baseline
  Fasting and 4 hour postprandial change in plasma inflammatory parameters including IL-1Ra and IL-1β (pg/mL by AlphaLISA)
Systemic inflammation | At 24 weeks
  Fasting and 4 hour postprandial change in plasma inflammatory parameters including IL-1Ra and IL-1β (pg/mL by AlphaLISA)
Disposition index | Baseline
  Calculated as glucose-induced insulin secretion (uU/mL/min) multiplied by insulin sensitivity (glucose infusion rate mg/kg/min) measured by Botnia clamp
Disposition index | At 24 weeks
  Calculated as glucose-induced insulin secretion (uU/mL/min) multiplied by insulin sensitivity (glucose infusion rate mg/kg/min) measured by Botnia clamp
Fatty acid profile in red blood cell phospholipid fraction | Baseline
  (As μmol/L by gas chromatography mass spectrometry)
Fatty acid profile in red blood cell phospholipid fraction | At 24 weeks
  (As μmol/L by gas chromatography mass spectrometry)
Body composition | Baseline
  Fat and lean body mass (as kg by dual energy x-ray absorptiometry)
Body composition | At 24 weeks
  Fat and lean body mass (as kg by dual energy x-ray absorptiometry)
Energy intake | Baseline
  (Average of 3 day energy intake as kcal/day collected by 3-day dietary records)
Energy intake | At 24 weeks
  (Average of 3 day energy intake as kcal/day collected by 3-day dietary records)
Physical activity | Baseline
  (using Godin Leisure Time Exercise Questionnaire)
Physical activity | At 24 weeks
  (using Godin Leisure Time Exercise Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: May Faraj, PDt, PhD, Principal Investigator — Montreal Clinical Research Institute/ University of Montreal
Locations (1):
- Montreal Clinical Research Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Frozen plasma and white adipose tissue samples (when sufficient) can be made available for analysis by other investigators. However data statistical analyses incorporating complete IPD must be conducted by the research team of Dr May Faraj as per subject consent form.

REFERENCES:
- [Background] Bissonnette S, Salem H, Wassef H, Saint-Pierre N, Tardif A, Baass A, Dufour R, Faraj M. Low density lipoprotein delays clearance of triglyceride-rich lipoprotein by human subcutaneous adipose tissue. J Lipid Res. 2013 May;54(5):1466-76. doi: 10.1194/jlr.P023176. Epub 2013 Feb 17. PMID 23417739
- [Background] Wassef H, Bissonnette S, Saint-Pierre N, Lamantia V, Cyr Y, Chretien M, Faraj M. The apoB-to-PCSK9 ratio: A new index for metabolic risk in humans. J Clin Lipidol. 2015 Sep-Oct;9(5):664-75. doi: 10.1016/j.jacl.2015.06.012. Epub 2015 Jul 2. PMID 26350813
- [Background] Lamantia V, Bissonnette S, Wassef H, Cyr Y, Baass A, Dufour R, Rabasa-Lhoret R, Faraj M. ApoB-lipoproteins and dysfunctional white adipose tissue: Relation to risk factors for type 2 diabetes in humans. J Clin Lipidol. 2017 Jan-Feb;11(1):34-45.e2. doi: 10.1016/j.jacl.2016.09.013. Epub 2016 Oct 3. PMID 28391908
- [Background] Skeldon AM, Faraj M, Saleh M. Caspases and inflammasomes in metabolic inflammation. Immunol Cell Biol. 2014 Apr;92(4):304-13. doi: 10.1038/icb.2014.5. Epub 2014 Feb 11. PMID 24518981
- [Background] Sattar N, Preiss D, Murray HM, Welsh P, Buckley BM, de Craen AJ, Seshasai SR, McMurray JJ, Freeman DJ, Jukema JW, Macfarlane PW, Packard CJ, Stott DJ, Westendorp RG, Shepherd J, Davis BR, Pressel SL, Marchioli R, Marfisi RM, Maggioni AP, Tavazzi L, Tognoni G, Kjekshus J, Pedersen TR, Cook TJ, Gotto AM, Clearfield MB, Downs JR, Nakamura H, Ohashi Y, Mizuno K, Ray KK, Ford I. Statins and risk of incident diabetes: a collaborative meta-analysis of randomised statin trials. Lancet. 2010 Feb 27;375(9716):735-42. doi: 10.1016/S0140-6736(09)61965-6. Epub 2010 Feb 16. PMID 20167359
- [Background] Ridker PM, Pradhan A, MacFadyen JG, Libby P, Glynn RJ. Cardiovascular benefits and diabetes risks of statin therapy in primary prevention: an analysis from the JUPITER trial. Lancet. 2012 Aug 11;380(9841):565-71. doi: 10.1016/S0140-6736(12)61190-8. PMID 22883507
- [Background] Lotta LA, Sharp SJ, Burgess S, Perry JRB, Stewart ID, Willems SM, Luan J, Ardanaz E, Arriola L, Balkau B, Boeing H, Deloukas P, Forouhi NG, Franks PW, Grioni S, Kaaks R, Key TJ, Navarro C, Nilsson PM, Overvad K, Palli D, Panico S, Quiros JR, Riboli E, Rolandsson O, Sacerdote C, Salamanca EC, Slimani N, Spijkerman AM, Tjonneland A, Tumino R, van der A DL, van der Schouw YT, McCarthy MI, Barroso I, O'Rahilly S, Savage DB, Sattar N, Langenberg C, Scott RA, Wareham NJ. Association Between Low-Density Lipoprotein Cholesterol-Lowering Genetic Variants and Risk of Type 2 Diabetes: A Meta-analysis. JAMA. 2016 Oct 4;316(13):1383-1391. doi: 10.1001/jama.2016.14568. PMID 27701660
- [Background] Schmidt AF, Swerdlow DI, Holmes MV, Patel RS, Fairhurst-Hunter Z, Lyall DM, Hartwig FP, Horta BL, Hypponen E, Power C, Moldovan M, van Iperen E, Hovingh GK, Demuth I, Norman K, Steinhagen-Thiessen E, Demuth J, Bertram L, Liu T, Coassin S, Willeit J, Kiechl S, Willeit K, Mason D, Wright J, Morris R, Wanamethee G, Whincup P, Ben-Shlomo Y, McLachlan S, Price JF, Kivimaki M, Welch C, Sanchez-Galvez A, Marques-Vidal P, Nicolaides A, Panayiotou AG, Onland-Moret NC, van der Schouw YT, Matullo G, Fiorito G, Guarrera S, Sacerdote C, Wareham NJ, Langenberg C, Scott R, Luan J, Bobak M, Malyutina S, Pajak A, Kubinova R, Tamosiunas A, Pikhart H, Husemoen LL, Grarup N, Pedersen O, Hansen T, Linneberg A, Simonsen KS, Cooper J, Humphries SE, Brilliant M, Kitchner T, Hakonarson H, Carrell DS, McCarty CA, Kirchner HL, Larson EB, Crosslin DR, de Andrade M, Roden DM, Denny JC, Carty C, Hancock S, Attia J, Holliday E, O'Donnell M, Yusuf S, Chong M, Pare G, van der Harst P, Said MA, Eppinga RN, Verweij N, Snieder H; LifeLines Cohort study group; Christen T, Mook-Kanamori DO, Gustafsson S, Lind L, Ingelsson E, Pazoki R, Franco O, Hofman A, Uitterlinden A, Dehghan A, Teumer A, Baumeister S, Dorr M, Lerch MM, Volker U, Volzke H, Ward J, Pell JP, Smith DJ, Meade T, Maitland-van der Zee AH, Baranova EV, Young R, Ford I, Campbell A, Padmanabhan S, Bots ML, Grobbee DE, Froguel P, Thuillier D, Balkau B, Bonnefond A, Cariou B, Smart M, Bao Y, Kumari M, Mahajan A, Ridker PM, Chasman DI, Reiner AP, Lange LA, Ritchie MD, Asselbergs FW, Casas JP, Keating BJ, Preiss D, Hingorani AD; UCLEB consortium; Sattar N. PCSK9 genetic variants and risk of type 2 diabetes: a mendelian randomisation study. Lancet Diabetes Endocrinol. 2017 Feb;5(2):97-105. doi: 10.1016/S2213-8587(16)30396-5. Epub 2016 Nov 29. PMID 27908689
- [Background] Ference BA, Robinson JG, Brook RD, Catapano AL, Chapman MJ, Neff DR, Voros S, Giugliano RP, Davey Smith G, Fazio S, Sabatine MS. Variation in PCSK9 and HMGCR and Risk of Cardiovascular Disease and Diabetes. N Engl J Med. 2016 Dec 1;375(22):2144-2153. doi: 10.1056/NEJMoa1604304. PMID 27959767
- [Background] Faraj M. LDL, LDL receptors, and PCSK9 as modulators of the risk for type 2 diabetes: a focus on white adipose tissue. J Biomed Res. 2020 Mar 12;34(4):251-259. doi: 10.7555/JBR.34.20190124. PMID 32701068
- [Background] Cyr Y, Bissonnette S, Lamantia V, Wassef H, Loizon E, Ngo Sock ET, Vidal H, Mayer G, Chretien M, Faraj M. White Adipose Tissue Surface Expression of LDLR and CD36 is Associated with Risk Factors for Type 2 Diabetes in Adults with Obesity. Obesity (Silver Spring). 2020 Dec;28(12):2357-2367. doi: 10.1002/oby.22985. Epub 2020 Oct 11. PMID 33043593
- [Background] Cyr Y, Lamantia V, Bissonnette S, Burnette M, Besse-Patin A, Demers A, Wabitsch M, Chretien M, Mayer G, Estall JL, Saleh M, Faraj M. Lower plasma PCSK9 in normocholesterolemic subjects is associated with upregulated adipose tissue surface-expression of LDLR and CD36 and NLRP3 inflammasome. Physiol Rep. 2021 Feb;9(3):e14721. doi: 10.14814/phy2.14721. PMID 33527668
- See also: IRCM website for recruitment — https://ircm.qc.ca/en/clinic/participate-in-a-clinical-study/study-aiming-reducing-risk-diabetes